CLINICAL TRIAL: NCT00067106
Title: Antiviral Therapy and HIV in the Genital Tract of Women
Brief Title: Antiviral Therapy and HIV in the Female Genital Tract
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Other Study IDs: AI04350
Record Dates: First submitted 2003-08-11; First posted 2003-08-13 (Estimated); Last update posted 2015-05-19 (Estimated); Status verified 2014-09

CONDITIONS: HIV Infections
Keywords: HIV; Women; Genital tract; Treatment experienced; Drug resistance
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood and genital tract collection
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: Women failing therapy: Participants will have study visits at study entry, 2 weeks after changing medications, then every 4 weeks until the amount of HIV in the blood and genital tract are undetectable. Drug levels in the blood and genital tract will also be measured at the first visit and after changing medications. Once the level of HIV is undetectable, women will be seen every 3 months for 36 months. Participants in Group 1 will be followed no more than 42 months.
- 2: Women suppressed on therapy: Participants will have study visits for blood and genital tract collections at study entry and then every 4 weeks for 12 months

SUMMARY:
HIV is found in both the blood and the genital tract. This study will compare the levels and types of HIV found in the blood with the levels and types of HIV found in the female genital tract.

Study hypotheses: 1) In the presence of antiretroviral therapy, viral replication within the female genital tract may lead to the development of drug resistance that is different from that of virus in the blood plasma. 2) Antiretroviral drug levels in the female genital tract may often be lower than in the blood plasma and differences in drug exposure may be associated with differences in virus replication and selection of resistant HIV variants during drug failure. 3) HIV can be recovered in vitro from cells in the female genital tract during successful therapy, and it may be genetically different from the HIV variants recovered from the blood cell latent reservoir on the same visit.

DETAILED DESCRIPTION:
Approximately 42 million adults are living with HIV/AIDS. The predominant mode of HIV transmission worldwide is through heterosexual contact. While many behavioral and biologic factors are associated with sexual transmission of HIV, viral load has been identified as the chief predictor of the risk of sexual transmission. Research has shown a strong correlation between blood plasma viral load and genital tract viral load. Antiretroviral medications can reduce blood plasma and genital tract HIV RNA levels, but antiretrovirals also lead to drug resistant HIV. In the United States and Europe, 2% to 27% of newly infected patients are infected with drug resistant HIV. There are reports of resistant genotypic variants in the genital tract that differ from variants found in the blood.

Understanding the dynamics of HIV in the genital tract is of great importance in strategies to control transmission of HIV. This study will evaluate the levels and variants of HIV in the blood and genital tracts of women taking antiretroviral medication.

Both women who are failing their current antiretroviral regimen (Group 1) and those who are fully suppressed on antiretroviral therapy (Group 2) will be enrolled in this study. Women in Group 1 will have study visits at study entry, 2 weeks after changing medications, then every 4 weeks until the amount of HIV in the blood and genital tract are undetectable. Drug levels in the blood and genital tract will also be measured at the first visit and after changing medications. Once the level of HIV is undetectable, women will be seen every 3 months for 36 months. Women in Group 1 will be followed no more than 42 months. Women in Group 2 will have study visits for blood and genital tract collections at study entry and then every 4 weeks for 12 months.

ELIGIBILITY:
Inclusion Criteria:

* HIV-infected
* Viral load below detectable limits for at least 6 months prior to study entry
* Have not failed an antiretroviral regimen or have failed only one previous antiretroviral regimen

Inclusion Criteria:

* HIV-infected
* Viral load more than 1,000 copies/ml on at least two occasions, with one viral load more than 10,000 copies/ml
* Expect to change to a new antiretroviral regimen

Exclusion Criteria:

Women not on antiretroviral therapy

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HIV-infected women who are failing their current antiretroviral regimen and those who are fully suppressed on antiretroviral therapy
Sampling Method: Non-Probability Sample
Enrollment: 130 (Actual)
Dates: Start 2003-07; Primary Completion 2007-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Antiviral Therapy and HIV in the Female Genital Tract | 2004-2009
  The primary analysis will be to compare resistance mutation patterns in blood plasma versus CVL population sequences.

SECONDARY OUTCOMES:
Antiviral Therapy and HIV in the Female Genital Tract | 2004-2009
  Compare resistance patterns in blood plasma versus endocervical sno-strip population sequences. Other secondary analyses will include comparison of resistance mutation patterns between blood and each of the other types of genital tract specimen. Comparisons across the 4 different genital tract specimen types will also be done. Phylogenies will be constructed to address whether there may be genetic differences between the blood and all genital tract specimen types in some subjects (aim 1a). The phylogenies will include blood and all genital tract specimen population sequences from each subject at the time of study entry.

CONTACTS AND LOCATIONS:
Overall Officials: Susan Cu-Uvin, MD, Principal Investigator — The Miriam Hospital, Brown Medical School
Locations (1):
- The Miriam Hospital, Providence, Rhode Island, United States

REFERENCES:
- [Result] Venkatesh KK, DeLong AK, Kantor R, Chapman S, Ingersoll J, Kurpewski J, De Pasquale MP, D'Aquila R, Caliendo AM, Cu-Uvin S. Persistent genital tract HIV-1 RNA shedding after change in treatment regimens in antiretroviral-experienced women with detectable plasma viral load. J Womens Health (Larchmt). 2013 Apr;22(4):330-8. doi: 10.1089/jwh.2012.3849. Epub 2013 Mar 26. PMID 23531097
- [Result] Cu-Uvin S, Caliendo AM. Genital tract HIV-1 RNA shedding among women with below detectable plasma viral load. AIDS. 2011 Mar 27;25(6):880-1. doi: 10.1097/QAD.0b013e328344ccf8. No abstract available. PMID 21412068
- [Result] Cu-Uvin S, DeLong AK, Venkatesh KK, Hogan JW, Ingersoll J, Kurpewski J, De Pasquale MP, D'Aquila R, Caliendo AM. Genital tract HIV-1 RNA shedding among women with below detectable plasma viral load. AIDS. 2010 Oct 23;24(16):2489-97. doi: 10.1097/QAD.0b013e32833e5043. PMID 20736815